CLINICAL TRIAL: NCT00348309
Title: A 54-week, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Effects of Rosiglitazone (Extended Release Tablets) as Adjunctive Therapy to Donepezil on Cognition and Overall Clinical Response in APOE ε4-stratified Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Rosiglitazone (Extended Release Tablets) As Adjunctive Therapy For Subjects With Mild To Moderate Alzheimer's Disease
Acronym: REFLECT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVA102672
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer's Disease
Keywords: apolipoprotein E; Alzheimer's disease; cognition; rosiglitazone; adjunctive therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Rosiglitazone Extended Release 2mg OD
  Interventions: Drug: Rosiglitazone Extended Release 2mg; Other: Donepezil
- Arm 2 (Experimental): Rosiglitazone Extended Release 8mg OD
  Interventions: Drug: Rosiglitazone Extended Release 8mg; Other: Donepezil
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo; Other: Donepezil

INTERVENTIONS:
Drug: Rosiglitazone Extended Release 2mg — Rosiglitazone Extended Release 2mg OD
  Arms: Arm 1
Drug: Rosiglitazone Extended Release 8mg — Rosiglitazone Extended Release 8mg OD
  Arms: Arm 2
Other: Placebo — Placebo
  Arms: Arm 3
Other: Donepezil — Donepezil (At least 6 months of ongoing donepezil therapy for Alzheimer's disease, with stable dosing for at least the last 2 months (and with no intent to change for the duration of the study).
  Other Names: Aricept

SUMMARY:
Rosiglitazone (RSG) has been tested in clinical studies and is approved by the FDA as a treatment for type II diabetes mellitus, a disease that occurs when the body is unable to effectively use glucose. RSG XR, the investigational drug used in this study, is an extended-release form of RSG.

This study tests whether RSG XR safely provides clinical benefit to people with mild to moderate Alzheimer's disease (AD) when combined with the currently approved AD medication, Aricept (donepezil). RSG XR is a new approach to AD therapy and this study tests a new way to treat AD by testing whether one's genetic makeup affects their response to the study drug. Clinical data suggesting that RSG may benefit AD patients was first seen in a small study performed at the University of Washington and then from a larger GSK study conducted in Europe and New Zealand. In the first study, subjects receiving RSG once daily for 6 months scored significantly better on 3 tests of memory and thought than those who did not receive RSG. In the GSK study, those that appeared to benefit most from treatment with RSG XR had a specific genetic pattern. They did not have the gene that caused them to produce the protein apolipoprotein E e4 (APOE e4). Subjects who have the APOE e4 gene may have two copies, one from each parent, or they may have only one APOE e4 gene meaning that they inherited either the APOE e2 or APOE e3 version of the gene, instead of APOE e4, from one of their parents. Subjects with one copy of the APOE e4 gene remained at their same level of thinking ability while those with two copies of the APOE e4 gene, continued to worsen during the 6-month treatment. The current study will more directly test the effectiveness or RSG XR on people who either have or lack the APOE e4 gene.

DETAILED DESCRIPTION:
A 54-week, double-blind, randomized, placebo-controlled, parallel-group study to investigate the effects of rosiglitazone (extended release tablets) as adjunctive therapy to donepezil on cognition and overall clinical response in APOE e4-stratified subjects with mild to moderate Alzheimer's disease (REFLECT-2)

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Male or female subject with a clinical diagnosis of probable Alzheimer's disease in accordance with NINCDS-ADRDA criteria.

(Note: National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and Alzheimer's Disease and Related Disorders Association (ADRDA).)

* Subject has mild to moderate Alzheimer's disease as defined by a MMSE score 10 to 26 inclusive at Screening.
* Hachinski Ischemia Score ≤ 4 at Screening.
* Age ≥50 and ≤90 years.
* At least 6 months of ongoing donepezil therapy for Alzheimer's disease, with stable dosing for at least the last 2 months (and with no intent to change for the duration of the study).
* Current use of medication is in accordance with the criteria listed in Table 2 (Permitted Medications,).
* Female subjects must be post-menopausal (i.e. >1 year without menstrual period), surgically sterile, or agree to use adequate method of contraception for the duration of the study. Female subjects who are pre-menopausal or who have been post-menopausal for <1 year must undertake pregnancy testing (urine test) at Visit 1, which must be negative.
* Brain CT or MRI scan performed within the past 12 months or at Screening, showing no evidence of any other potential cause of dementia other than Alzheimer's disease.

(Note: Questionable CT or MRI scans should be discussed with the medical monitor, using central imaging guidelines.)

* Neurological exam without focal changes (excluding changes attributable to AD or peripheral trauma).
* Subject has the ability to comply with procedures for cognitive and other testing.
* Subject lives with (or has substantial periods of contact with) a regular caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status.

Note: A non-cohabiting caregiver must spend sufficient time with the subject so that, in the opinion of the Investigator, the caregiver can reliably assess cognitive function, activities and behavior, and report on the subject's compliance and health. As caregiver time spent with a potential subject is anticipated to be highly variable across countries and cultures, GSK will consider a variety of different measures by which this stipulation may be met, and GSK should be consulted if adequacy of a caregiver situation is in doubt. However, as guidance, the ability for a caregiver to meet his/her expected responsibilities for this study would normally be possible when the caregiver spends no less than 10 hours per week with the subject, divided over multiple days.)

* Subject has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative.

(Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations and ethics committee policy.)

* Caregiver has provided full written informed consent on his/her own behalf prior to the performance of any protocol-specified procedure.
* Subjects considered for enrolment must have a QTc (either QTc B (Bazett's correction) or QTc F (Fridericia's correction)) <450msec at Visit 1, with the exception of subjects with bundle branch block (for whom either QTc B or QTc F must be <480msec).
* (Note: For the purposes of these criteria, QTc B is defined as (QT interval [msec]) / (square root of RR interval [seconds]); and QTc F is defined as (QT interval [msec]) / (cube root of RR interval [seconds]).)

Exclusion criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Diagnosis of possible, probable, or definite vascular dementia in accordance with NINDS-AIREN criteria.

(Note: National Institute of Neurological Disorders and Stroke (NINDS) and Association Internationale pour la Recherche et l'Enseignement en Neurosciences (AIREN).)

* History or evidence of any other CNS disorder that could be interpreted as a cause of dementia: e.g. cerebrovascular disease (stroke, hemorrhage), structural abnormality, epilepsy, infectious or inflammatory/demyelinating CNS conditions, Parkinson's disease.
* Evidence of the following disorders: current vitamin B12 deficiency, positive syphilis serology, or active thyroid dysfunction (particularly that suggestive of hypothyroidism), including abnormally high or low serum levels of thyroid stimulating hormone (TSH) that are clinically significant in the opinion of the investigator.

(Note: Testing is required for each parameter only when no result is available from previous 12 months.)

* History of Type 1 diabetes mellitus or secondary diabetes mellitus.
* Type 2 diabetes mellitus where the subject is being treated with insulin, a PPARγ agonist, or an insulin secretagogue (e.g. a sulfonylurea or glitinide).
* Any patient with an HbA1c ≥8.5%. (See Section 6.3.7.4 for Safety Measures for Enrolled Subjects with Type 2 Diabetes Mellitus.)
* History or clinical/investigational evidence of congestive heart failure defined by the New York Heart Association criteria (Class I to IV cardiac status;).
* History of cardiovascular event within the last 6 months (i.e. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia; or major intervention (e.g. cardiac surgery or angiography plus stenting) scheduled).
* History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study, major depressive disorder (according to DSM-IV) in the past year, or current active depression requiring initiation of treatment.

(Note: If not currently treated, but active depression is suspected, the Cornell Scale for Depression in Dementia (CSDD) can be used by the Investigator as a guide for deciding whether a prospective subject requires treatment. If the subject has a CSDD score >7, the Investigator should decide if the subject has depression in need of prescribed medication, and a CSDD >12 is considered a strong indicator that treatment is needed. Subjects will be allowed to re-screen after their depression has been adequately managed for >3 months.)

* History or presence of gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or any other clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* Clinically significant peripheral edema at the time of screening.
* Current or recent drug or alcohol abuse or dependence (defined by DSM-IV criteria for substance-related disorders), or recent or remote history of the same if that could be a contributing factor to the dementia.
* Systolic blood pressure >165 or <90 mmHg or diastolic blood pressure >95 or <60 mmHg at the time of screening.
* Clinically significant anemia (i.e. hemoglobin <11 g/dL for males or <10 g/dL for females) or presence of hemoglobinopathies which would prevent accurate assessment of HbA1c.
* Abnormal kidney function tests (>1.5 the upper limit of normal (ULN)).
* ALT, AST, or alkaline phosphatase values >2.5 times the ULN, total bilirubin values >1.5 times the ULN, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C).

(Note: For subjects with a diagnosis of Gilberts Syndrome and an isolated increase in total bilirubin >1.5 ULN, fractionation should be performed. If all of the following conditions are met, the patient may enter or remain in the study, even if total bilirubin >1.5 ULN:

* an elevated unconjugated (indirect) bilirubin;
* the percentage of direct bilirubin <35%;
* ALT, AST, and alkaline phosphatase <2.5 ULN if subject is in screening (<2.0 ULN for Canadian subjects only), or ≤3 ULN if subject is already randomized into the study)
* History of a bone marrow transplant.
* Subject is unable (with assistance, if appropriate) to take study medication as prescribed throughout the study or is at risk of non-compliance with study medication or procedures.
* Subject is an immediate family member or employee of the participating Investigator, of any of the participating site staff, or of GSK.
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.
* The French subject has participated in any study using an investigational drug during the previous 30 days or 5 half-lives (whichever is longer).
* Cognitive tasks prescribed for cognitive rehabilitation and performed under medical supervision are prohibited for 6 months prior to Screening, as well as for the duration of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1496 (Actual)
Dates: Start 2006-07-06; Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (203):
- United States (39):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Nutley, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, South Ogden, Utah
  - GSK Investigational Site, Bennington, Vermont
- Argentina (6):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Austria (3):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Ribeirão Preto
  - GSK Investigational Site, São Paulo
- Canada (15):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Medicine Hat, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Whitby, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Québec
- Chile (4):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Czechia (2):
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
- France (29):
  - GSK Investigational Site, Angoulême
  - GSK Investigational Site, Arcachon
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Bourg-en-Bresse
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Issy-les-Moulineaux
  - GSK Investigational Site, Ivry
  - GSK Investigational Site, Luynes
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rodez
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Jean-de-Luz
  - GSK Investigational Site, Saint-Nicolas-de-Port
  - GSK Investigational Site, Saint-Ouen-la-Rouërie
  - GSK Investigational Site, Tinténiac
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Verny
  - GSK Investigational Site, Vichy
- Germany (33):
  - GSK Investigational Site, Böblingen, Baden-Wurttemberg
  - GSK Investigational Site, Ostfildern, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuburg an der Donau, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Bockhorn, Lower Saxony
  - GSK Investigational Site, Ganderkesee, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bad Honnef, North Rhine-Westphalia
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Jülich, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Remscheid, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Hamburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Szeged
- India (7):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Varanasi
- Italy (15):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, San Felice A Cancello Caserta, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Rho, Lombardy
  - GSK Investigational Site, Ancona, The Marches
  - GSK Investigational Site, Arezzo, Tuscany
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Verona, Veneto
- Japan (15):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Mexico (3):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- Poland (7):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Mosina
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Warsaw
- Portugal (2):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
- Spain (13):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Harrington C, Sawchak S, Chiang C, Davies J, Donovan C, Saunders AM, Irizarry M, Jeter B, Zvartau-Hind M, van Dyck CH, Gold M. Rosiglitazone does not improve cognition or global function when used as adjunctive therapy to AChE inhibitors in mild-to-moderate Alzheimer's disease: two phase 3 studies. Curr Alzheimer Res. 2011 Aug;8(5):592-606. doi: 10.2174/156720511796391935. PMID 21592048
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVA102672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on participants with mild to moderate Alzheimer's disease(AD), who received donepezil for at least 6 months and who received a stable dose of donepezil for at least 2 months immediately before study entry from 06 July 2006 to 28 January 2009 across 228 centers of 19 countries.
Pre-assignment Details: A total of 1496 participants were randomized for the study, out of which seventeen participants did not receive study medication. A total of 1479 were included in the Safety population.
Groups:
- Placebo: Participants received rosiglitazone extended release matching placebo tablet orally, once daily until Week 54.
- 2mg Rosiglitazone Extended Release: Participants received rosiglitazone extended release 2 milligram (mg) tablet orally, once daily until Week 48 followed by placebo tablet orally once daily until Week 54.
- 8mg Rosiglitazone Extended Release: Participants received rosiglitazone extended release 4 mg tablet orally, once daily until Week 4 followed by 8 mg tablet orally once daily from Week 4 until Week 48 followed by placebo tablet orally once daily until Week 54.
Period: Overall Study
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Started | 496 | 494 | 489
Completed | 362 | 396 | 346
Not Completed | 134 | 98 | 143
Not completed — Adverse Event | 56 | 28 | 63
Not completed — Lost to Follow-up | 6 | 7 | 4
Not completed — Protocol Violation | 7 | 12 | 7
Not completed — Withdrawal by Subject | 33 | 37 | 40
Not completed — Non-compliance | 8 | 6 | 8
Not completed — Death of caregiver | 1 | 0 | 1
Not completed — Lack of insight, dementia | 1 | 0 | 0
Not completed — Wrong bottle allocated | 1 | 0 | 0
Not completed — Caregiver sick | 1 | 0 | 0
Not completed — Use of prohibited medication | 5 | 2 | 2
Not completed — Caregiver withdrawal | 3 | 0 | 7
Not completed — Unable to complete ET visit | 1 | 0 | 0
Not completed — PI closing medical practice | 1 | 0 | 0
Not completed — Principal investigator's decision | 1 | 0 | 0
Not completed — No disponibility of medication | 1 | 0 | 0
Not completed — Worsened neurodegenerative disease | 1 | 0 | 0
Not completed — Cognitive and behaviour worsening | 2 | 0 | 0
Not completed — Worsening of alzheimer | 1 | 0 | 1
Not completed — Did not appear in time for Visit 3 | 1 | 0 | 0
Not completed — Participant died | 2 | 1 | 1
Not completed — Decision of sponsor | 1 | 0 | 0
Not completed — Ineffectiveness of treatment | 0 | 1 | 0
Not completed — A foul of exclusion criteria | 0 | 1 | 0
Not completed — Participant was hospitalized | 0 | 1 | 0
Not completed — Sponsor refuseal | 0 | 1 | 1
Not completed — Forgot often medication | 0 | 1 | 0
Not completed — Medical Monitor decision | 0 | 0 | 1
Not completed — Increased dose of Aricept | 0 | 0 | 1
Not completed — Site closure | 0 | 0 | 1
Not completed — Adverse event not attended | 0 | 0 | 1
Not completed — ECG abnormal | 0 | 0 | 2
Not completed — Cardiologist recommendations | 0 | 0 | 1
Not completed — HCV career | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release | Total
Number analyzed (Participants) | 496 | 494 | 489 | 1479
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.2 (7.95) | 74.5 (8.06) | 74.4 (7.83) | 74.4 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 286 | 305 | 895
  Male | 192 | 208 | 184 | 584
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 97 | 86 | 82 | 265
  Not Hispanic or Latino | 399 | 408 | 407 | 1214

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Total Score at Week 48
Description: ADAS is a performance-based test that measures specific cognitive and behavioral dysfunctions in participants with Alzheimer's Disease. The cognitive subscale of the ADAS (ADAS-Cog) comprises 11 items that are summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. Change from baseline is calculated as Week 48 value minus the baseline value. APOE4 negative, All except E4/E4's: comprised of APOE4 negative and E4 heterozygote and full population was analyzed for this outcome measure. A hierarchical testing procedure was used to control for the two rosiglitazone dose groups and the genetic subgroups. Least square mean is entered for adjusted mean.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population included all the participants who were randomized to treatment, who had received at least one dose of study medication and who had at least one post baseline efficacy assessment. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  APOE4 negatives: number analyzed (Participants) | 153 | 172 | 141
  APOE4 negatives | 2.9 (0.54) | 1.6 (0.42) | 2.7 (0.56)
  All except E4/E4s: number analyzed (Participants) | 317 | 350 | 285
  All except E4/E4s | 3.1 (0.36) | 2.1 (0.29) | 3.1 (0.37)
  Full populations: number analyzed (Participants) | 356 | 391 | 333
  Full populations | 3.4 (0.35) | 2.4 (0.30) | 3.2 (0.35)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis — APOE4 negatives; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.7 to -0.0]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.808, Mixed Models Analysis — APOE4 negatives; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.7 to 1.3]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis — All except E4/E4s; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.9 to -0.1]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis — All except E4/E4s; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis — Full population; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.9 to -0.2]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.661, Mixed Models Analysis — Full population; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.2 to 0.7]

2. Primary Outcome: Change From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) at Week 48 for APOE E4
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Change from baseline is calculated as Week 48 value minus the baseline value. APOE4 negative, All except E4/E4's: comprised of APOE4 negative and E4 heterozygote and full population was analyzed for this outcome measure. A hierarchical testing procedure was used to control for the two rosiglitazone dose groups and the genetic subgroups.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- 2mg Rosiglitazone Extended Release: Participants received rosiglitazone extended release 2 mg tablet orally, once daily until Week 48 followed by placebo tablet orally once daily until Week 54.
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  APOE4 negatives: number analyzed (Participants) | 146 | 169 | 139
  APOE4 negatives | 1.3 (0.21) | 0.8 (0.16) | 1.5 (0.20)
  All except E4/E4s: number analyzed (Participants) | 309 | 343 | 283
  All except E4/E4s | 1.5 (0.14) | 1.0 (0.12) | 1.7 (0.14)
  Full population: number analyzed (Participants) | 347 | 384 | 331
  Full population | 1.6 (0.14) | 1.0 (0.12) | 1.7 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis — APOE4 negatives; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.587, Mixed Models Analysis — APOE4 negatives; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — All except E4/E4s; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.402, Mixed Models Analysis — All except E4/E4s; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Full population; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.478, Mixed Models Analysis — Full population; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.5]

3. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia Scale (DAD) Total Score
Description: The DAD measures instrumental and basic activities of daily living in participants with Alzheimer's Disease (AD). This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. The scale includes 23 items relating to instrumental activities of daily living and 17 items relating to basic self-care. Each item can be scored as 1 = yes, 0 = no, non applicable = NA. Total score was obtained by adding the rating for each question and converting this total score out of 100. The total score ranged from 0 to 100, where higher score indicated better function and lower score indicated greater severity of symptoms; a positive change from baseline indicated an improvement. Change from baseline is calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 8, 16, 24 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 436 | 458 | 441
Scores on a scale
  At Week 8 | 0.1 (0.56) | -0.5 (0.48) | -1.1 (0.47)
  At Week 16 | -1.6 (0.62) | -1.6 (0.59) | -2.1 (0.56)
  At Week 24 | -3.5 (0.69) | -2.2 (0.64) | -3.3 (0.69)
  At Week 48 | -7.8 (0.82) | -5.7 (0.78) | -8.4 (0.84)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.340, Mixed Models Analysis — Week 8; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.0 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — Week 8; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.5 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.910, Mixed Models Analysis — Week 16; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.7 to 1.5]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.521, Mixed Models Analysis — Week 16; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.1 to 1.0]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.154, Mixed Models Analysis — Week 24; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.5 to 3.0]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.836, Mixed Models Analysis — Week 24; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.6 to 2.0]
Statistical Analysis 7: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.1 to 4.2]
Statistical Analysis 8: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.566, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.9 to 1.6]

4. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing).The NPI Psychosis Subscale consists of the two domains of Delusions and Hallucinations, calculated by adding the Individual Item Scores, to yield a possible total score of 0 to 24. Lower score=less severity. Change from baseline is calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 8, 16, 24 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  At Week 8: number analyzed (Participants) | 440 | 458 | 442
  At Week 8 | -0.3 (0.39) | -0.7 (0.32) | -0.3 (0.39)
  At Week 16: number analyzed (Participants) | 425 | 442 | 415
  At Week 16 | -0.3 (0.43) | -0.6 (0.36) | 0.1 (0.43)
  At Week 24: number analyzed (Participants) | 411 | 425 | 390
  At Week 24 | 0.4 (0.47) | -0.2 (0.39) | 0.2 (0.48)
  At Week 48: number analyzed (Participants) | 359 | 395 | 345
  At Week 48 | 1.6 (0.61) | 0.1 (0.44) | 1.8 (0.55)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.414, Mixed Models Analysis — Week 8; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.3 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.931, Mixed Models Analysis — Week 8; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 1.1]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.485, Mixed Models Analysis — Week 16; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.4 to 0.7]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.550, Mixed Models Analysis — Week 16; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.8 to 1.5]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis — Week 24; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.5]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.732, Mixed Models Analysis — Week 24; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.5 to 1.0]
Statistical Analysis 7: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.9 to -0.0]
Statistical Analysis 8: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.4 to 1.8]

5. Secondary Outcome: Change From Screening in Mini Mental State Examination (MMSE) Total Score
Description: The MMSE consists of 11 tests of orientation, memory (recent and immediate), concentration, language and praxis. The scale was completed by the investigator, based on the performance of the participant, and took approximately 5 to 10 minutes to administer. The scores from 11 tests were combined to obtain the total score. The total scores range from 0 to 30, with lower scores indicating greater cognitive impairment and higher score indicating better outcome; a positive change from screening indicated an improvement. The total MMSE score for participants at screening was between 10 and 26, inclusive, in order to be eligible to participate in the trial. Change from screening is calculated as endpoint value minus the screening value.
Time Frame: Screening (Week -4) and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 348 | 388 | 335
Score on a scale | -1.6 (0.21) | -1.6 (0.20) | -1.7 (0.21)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.870, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.617, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4]

6. Secondary Outcome: Change From Baseline in the Domains of the Resource Utilization in Dementia Scale (RUD)
Description: The RUD instrument was developed as a comprehensive tool to assess the amount of resource use among demented patients. RUD assessd both formal and informal resource use of the patient and the primary caregiver, making it possible to calculate costs from a societal perspective. Q1 corresponds to the number of hours during the last month the caregiver spent assisting the patient with toilet visits, eating, dressing, grooming, walking and bathing and Q2 corresponds to the number of hours during the last month the caregiver spent assisting the patient with shopping, food preparation, housekeeping, laundry, transportation, taking medication and managing financial matters. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented.
Time Frame: Baseline (Week 0), Week 12, 24, 36 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
hours
  Q1: Week 12: number analyzed (Participants) | 386 | 408 | 379
  Q1: Week 12 | 1.6 (2.25) | 2.4 (2.50) | -0.1 (3.18)
  Q1: Week 24: number analyzed (Participants) | 386 | 380 | 347
  Q1: Week 24 | 10.7 (3.52) | 3.4 (1.84) | 7.0 (4.06)
  Q1: Week 36: number analyzed (Participants) | 342 | 361 | 327
  Q1: Week 36 | 16.3 (3.60) | 10.0 (3.43) | 15.2 (4.95)
  Q1: Week 48: number analyzed (Participants) | 320 | 351 | 310
  Q1: Week 48 | 21.7 (4.16) | 17.0 (4.17) | 18.1 (4.72)
  Q2: Week 12: number analyzed (Participants) | 171 | 183 | 162
  Q2: Week 12 | -6.4 (4.64) | 2.4 (4.16) | 1.5 (4.50)
  Q2: Week 24: number analyzed (Participants) | 162 | 170 | 150
  Q2: Week 24 | 0.3 (4.89) | 1.6 (4.17) | 6.5 (4.88)
  Q2: Week 36: number analyzed (Participants) | 153 | 162 | 141
  Q2: Week 36 | 5.0 (5.34) | 4.6 (4.44) | 13.3 (5.35)
  Q2: Week 48: number analyzed (Participants) | 139 | 157 | 137
  Q2: Week 48 | 10.8 (5.51) | 8.4 (4.88) | 27.0 (6.24)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Week 12 Q1; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-5.2 to 6.9]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.643, Mixed Models Analysis — Week 12Q1; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-9.0 to 5.6]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.052, Mixed Models Analysis — Week 24 Q1; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-14.7 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.481, Mixed Models Analysis — Week 24 Q1; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-14.0 to 6.6]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.195, Mixed Models Analysis — Week 36 Q1; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-15.6 to 3.2]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.857, Mixed Models Analysis — Week 36 Q1; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-12.9 to 10.7]
Statistical Analysis 7: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.422, Mixed Models Analysis — Week 48 Q1; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-15.9 to 6.7]
Statistical Analysis 8: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.562, Mixed Models Analysis — Week 48 Q1; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-15.7 to 8.6]
Statistical Analysis 9: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.129, Mixed Models Analysis — Week 12 Q2; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [-2.6 to 20.2]
Statistical Analysis 10: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.194, Mixed Models Analysis — Week 12 Q2; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [-4.0 to 19.9]
Statistical Analysis 11: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.832, Mixed Models Analysis — Week 24 Q2; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-10.5 to 13.1]
Statistical Analysis 12: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.351, Mixed Models Analysis — Week 24 Q2; Mean Difference (Final Values) = 6.1, 95% CI 2-sided [-6.8 to 19.1]
Statistical Analysis 13: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.949, Mixed Models Analysis — Week 36 Q2; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-13.3 to 12.5]
Statistical Analysis 14: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.253, Mixed Models Analysis — Week 36 Q2; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [-6.0 to 22.6]
Statistical Analysis 15: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.735, Mixed Models Analysis — Week 48 Q2; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-16.2 to 11.4]
Statistical Analysis 16: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.046, Mixed Models Analysis — Week 48 Q2; Mean Difference (Final Values) = 16.2, 95% CI 2-sided [0.3 to 32.0]

7. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Proxy Version (EQ-5D Proxy) Scale Total Score Assessed by Thermometer (Visual Analog Scale [VAS]) and Utility
Description: The EQ-5D Proxy is a two part scale that evaluated the participant's health status via Thermometer and Utility scores. The Thermometer score was the caregiver's rating of the participant's overall health status on a VAS (0 ["worst possible status"] to 100 ["best imaginable status"]). The Utility score was a caregiver rating of health status on dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression] where '1' indicated better health state (no problems); '3' indicated worst health state ("confined to bed"). Total possible score was the sum of individual items, ranged from 5 to 15; lower score indicated a better health state and higher score indicated greater severity of symptoms. A positive change from baseline indicated improvement in the Thermometer score and a negative change from baseline indicated improvement in the Utility score. Change from baseline is calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 12, 36 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  Thermometer: Week 12: number analyzed (Participants) | 425 | 449 | 413
  Thermometer: Week 12 | 0.5 (0.84) | 0.3 (0.82) | -0.5 (0.94)
  Thermometer: Week 36: number analyzed (Participants) | 381 | 404 | 362
  Thermometer: Week 36 | 0.8 (0.95) | -1.6 (0.97) | -2.1 (1.03)
  Thermometer: Week 48: number analyzed (Participants) | 352 | 389 | 337
  Thermometer: Week 48 | -1.5 (1.05) | -0.3 (0.96) | -2.4 (1.08)
  Utility: Week 12: number analyzed (Participants) | 425 | 448 | 414
  Utility: Week 12 | 0.01 (0.009) | 0.02 (0.009) | -0.01 (0.010)
  Utility: Week 36: number analyzed (Participants) | 381 | 403 | 363
  Utility: Week 36 | -0.02 (0.011) | -0.01 (0.010) | -0.04 (0.012)
  Utility: Week 48: number analyzed (Participants) | 351 | 389 | 337
  Utility: Week 48 | -0.04 (0.012) | -0.02 (0.011) | -0.05 (0.013)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.914, Mixed Models Analysis — Week 12 Thermometer; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.3 to 2.0]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.415, Mixed Models Analysis — Week 12 Thermometer; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.3 to 1.4]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis — Week 36 Thermometer; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.9 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — Week 36 Thermometer; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.6 to -0.3]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.392, Mixed Models Analysis — Week 48 Thermometer; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.5 to 3.8]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.557, Mixed Models Analysis — Week 48 Thermometer; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.7 to 2.0]
Statistical Analysis 7: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.320, Mixed Models Analysis — Week 12 Utility; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 8: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.180, Mixed Models Analysis — Week 12 Utility; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.04 to 0.01]
Statistical Analysis 9: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.498, Mixed Models Analysis — Week 36 Utility; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.02 to 0.04]
Statistical Analysis 10: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis — Week 36 Utility; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.06 to 0.00]
Statistical Analysis 11: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis — Week 48 Utility; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.00 to 0.06]
Statistical Analysis 12: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.640, Mixed Models Analysis — Week 48 Utility; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.04 to 0.03]

8. Secondary Outcome: Change From Baseline in ADAS-Cog Total Score for Observed Cases at Weeks 8, 16, 24, 36 and 48
Description: ADAS is a performance-based test that measures specific cognitive and behavioral dysfunctions in patients with Alzheimer's Disease. The cognitive subscale of the ADAS (ADAS-Cog) comprises 11 items that are summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. Change from baseline is calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 36 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  Week 8: number analyzed (Participants) | 435 | 457 | 437
  Week 8 | -0.2 (4.21) | -0.6 (4.57) | -0.2 (4.44)
  Week 16: number analyzed (Participants) | 422 | 441 | 411
  Week 16 | -0.1 (5.09) | -0.5 (4.76) | 0.1 (5.13)
  Week 24: number analyzed (Participants) | 404 | 425 | 386
  Week 24 | 1.0 (5.86) | -0.2 (5.17) | 0.8 (5.66)
  Week 36: number analyzed (Participants) | 378 | 402 | 362
  Week 36 | 1.8 (6.08) | 1.3 (5.79) | 2.2 (6.40)
  Week 48: number analyzed (Participants) | 358 | 393 | 333
  Week 48 | 2.9 (6.85) | 2.1 (6.25) | 2.6 (6.76)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.105, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.6 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.483, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.6]

9. Secondary Outcome: Change From Baseline in CDR-SB Score for Observed Cases at Weeks 12, 24, 36 and 48
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Change from baseline is calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 12, 24, 36 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  Week 12: number analyzed (Participants) | 423 | 446 | 414
  Week 12 | 0.4 (1.55) | 0.3 (1.36) | 0.3 (1.40)
  Week 24: number analyzed (Participants) | 402 | 421 | 382
  Week 24 | 0.7 (2.01) | 0.5 (1.67) | 0.8 (1.83)
  Week 36: number analyzed (Participants) | 374 | 400 | 357
  Week 36 | 1.0 (2.26) | 0.7 (2.06) | 1.2 (2.30)
  Week 48: number analyzed (Participants) | 349 | 385 | 331
  Week 48 | 1.5 (2.68) | 1.0 (2.28) | 1.6 (2.56)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.554, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.5]

10. Secondary Outcome: Change in ADAS-Cog Total Score for Observed Cases at Week 54 Compared to Week 48
Description: ADAS is a performance-based test that measures specific cognitive and behavioral dysfunctions in patients with Alzheimer's Disease. The cognitive subscale of the ADAS (ADAS-Cog) comprises 11 items that are summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. Change was calculated as endpoint value (Week 54) minus Week 48 value.
Time Frame: Week 48 and 54
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 332 | 366 | 305
Score on a scale | 0.7 (0.28) | 1.1 (0.27) | 1.1 (0.29)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.292, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.1]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.297, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.1]

11. Secondary Outcome: Change in CDR-SB Total Score at Week 54 Compared to Week 48
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. Change was calculated as endpoint value (Week 54) minus Week 48 value.
Time Frame: Week 48 and 54
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 328 | 364 | 302
Score on a scale | 0.2 (0.07) | 0.2 (0.07) | 0.1 (0.07)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.598, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.073, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0]

12. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 48
Description: Blood samples of participants were collected for HbA1c assessment. HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Change from Baseline in HbA1c was calculated as the value at Week 48 minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of total hemoglobin
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 321 | 352 | 313
Percentage of total hemoglobin | 0.14 (0.020) | 0.21 (0.020) | 0.18 (0.020)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.02 to 0.12]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.140, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.01 to 0.09]

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. The data was reported for prospective period.
Time Frame: Up to Week 54
Population: The safety population included all participants randomized to treatment and received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 496 | 494 | 489
Participants
  Any TEAEs | 304 | 273 | 327
  Any SAEs | 62 | 45 | 50

14. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure (BP)
Description: The plethysmographic method was used to measure BP throughout the study. Change in Systolic and Diastolic BP was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 4, 8, 12, 16, 24, 36, 48 and 56
Population: Safety population. Only those participants available at the specified time points were analyzed. Data for Site 040449 was not included in analysis due to audit finding.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 477 | 481 | 470
Millimeter of mercury (mmHg)
  Systolic BP Week 4: number analyzed (Participants) | 457 | 469 | 457
  Systolic BP Week 4 | -0.7 (15.21) | -1.0 (13.21) | -2.3 (13.43)
  Systolic BP Week 8: number analyzed (Participants) | 436 | 460 | 434
  Systolic BP Week 8 | -0.3 (15.49) | -0.7 (14.55) | -2.9 (14.49)
  Systolic BP Week 12: number analyzed (Participants) | 431 | 454 | 415
  Systolic BP Week 12 | -0.5 (16.48) | -2.5 (14.49) | -4.2 (15.25)
  Systolic BP Week 16: number analyzed (Participants) | 425 | 442 | 411
  Systolic BP Week 16 | -0.8 (15.80) | -1.7 (14.80) | -3.7 (15.75)
  Systolic BP Week 24: number analyzed (Participants) | 413 | 431 | 392
  Systolic BP Week 24 | -1.2 (15.95) | -1.0 (15.22) | -3.5 (14.74)
  Systolic BP Week 36: number analyzed (Participants) | 384 | 406 | 367
  Systolic BP Week 36 | -1.6 (16.65) | -0.3 (15.79) | -2.7 (15.97)
  Systolic BP Week 48: number analyzed (Participants) | 363 | 397 | 345
  Systolic BP Week 48 | -1.0 (17.08) | -0.6 (15.05) | -2.5 (16.55)
  Systolic BP Week 54: number analyzed (Participants) | 345 | 385 | 321
  Systolic BP Week 54 | 0.0 (17.24) | -1.1 (14.95) | -2.3 (15.56)
  Diastolic BP Week 4: number analyzed (Participants) | 457 | 469 | 457
  Diastolic BP Week 4 | -0.4 (9.54) | -0.7 (9.21) | -1.2 (8.51)
  Diastolic BP Week 8: number analyzed (Participants) | 436 | 460 | 434
  Diastolic BP Week 8 | -0.0 (9.55) | -0.9 (9.20) | -2.1 (9.21)
  Diastolic BP Week 12: number analyzed (Participants) | 431 | 454 | 415
  Diastolic BP Week 12 | 0.0 (9.63) | -1.3 (9.25) | -2.5 (9.49)
  Diastolic BP Week 16: number analyzed (Participants) | 425 | 442 | 411
  Diastolic BP Week 16 | -0.7 (9.78) | -1.3 (9.16) | -3.0 (9.62)
  Diastolic BP Week 24: number analyzed (Participants) | 413 | 431 | 392
  Diastolic BP Week 24 | -1.1 (9.87) | -1.2 (9.55) | -2.6 (9.48)
  Diastolic BP Week 36: number analyzed (Participants) | 384 | 406 | 367
  Diastolic BP Week 36 | -1.2 (10.27) | -0.6 (9.94) | -3.3 (10.68)
  Diastolic BP Week 48: number analyzed (Participants) | 363 | 397 | 345
  Diastolic BP Week 48 | -0.8 (10.85) | -0.5 (10.02) | -1.9 (11.07)
  Diastolic BP Week 54: number analyzed (Participants) | 345 | 385 | 321
  Diastolic BP Week 54 | -0.9 (10.35) | -0.4 (9.62) | -1.8 (10.04)

15. Secondary Outcome: Mean Change From Baseline in Heart Rate
Description: Mean Change From Baseline in heart rate was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 4, 8, 12, 16, 24, 36, 48 and 56
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: beats per min (bpm)
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 477 | 481 | 470
beats per min (bpm)
  Week 4: number analyzed (Participants) | 457 | 468 | 457
  Week 4 | 0.8 (8.42) | 1.1 (7.95) | 0.6 (8.36)
  Week 8: number analyzed (Participants) | 435 | 459 | 434
  Week 8 | 1.5 (8.98) | 1.3 (9.19) | 1.0 (8.91)
  Week 12: number analyzed (Participants) | 430 | 453 | 414
  Week 12 | 1.6 (9.06) | 1.8 (9.04) | 0.7 (9.68)
  Week 16: number analyzed (Participants) | 425 | 441 | 411
  Week 16 | 1.0 (9.23) | 1.3 (9.18) | 0.8 (9.52)
  Week 24: number analyzed (Participants) | 413 | 431 | 392
  Week 24 | 0.9 (9.41) | 1.3 (8.70) | 0.8 (10.19)
  Week 36: number analyzed (Participants) | 382 | 406 | 367
  Week 36 | 0.9 (9.30) | 1.8 (9.42) | 1.1 (9.58)
  Week 48: number analyzed (Participants) | 361 | 397 | 344
  Week 48 | 1.2 (9.10) | 1.4 (8.92) | 0.7 (9.43)
  Week 54: number analyzed (Participants) | 344 | 384 | 321
  Week 54 | 0.5 (10.10) | 1.4 (9.55) | 0.0 (11.05)

16. Secondary Outcome: Mean Change From Baseline in Weight
Description: Body weight was measured at all visits, without shoes and wearing light clothing. Mean Change From Baseline in Weight was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 4, 8, 12, 16, 24, 36, 48 and 56
Population: Safety population. Here, n=number of participants with observed data contributing to the analysis. Data for Site 040449 was not included in analysis due to audit finding.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 477 | 481 | 470
kilogram (kg)
  Week 4: number analyzed (Participants) | 456 | 471 | 458
  Week 4 | 0.1 (2.04) | 0.2 (1.66) | 0.3 (1.88)
  Week 8: number analyzed (Participants) | 436 | 460 | 435
  Week 8 | 0.2 (2.35) | 0.3 (1.95) | 0.7 (2.37)
  Week 12: number analyzed (Participants) | 430 | 453 | 414
  Week 12 | 0.2 (2.50) | 0.3 (2.09) | 0.9 (2.33)
  Week 16: number analyzed (Participants) | 425 | 441 | 412
  Week 16 | 0.1 (2.88) | 0.3 (2.44) | 1.0 (2.56)
  Week 24: number analyzed (Participants) | 413 | 430 | 391
  Week 24 | 0.1 (2.88) | 0.6 (2.77) | 0.9 (3.26)
  Week 36: number analyzed (Participants) | 384 | 405 | 367
  Week 36 | 0.0 (3.37) | 0.7 (3.00) | 1.3 (3.92)
  Week 48: number analyzed (Participants) | 363 | 396 | 346
  Week 48 | 0.4 (3.54) | 0.8 (3.47) | 1.3 (4.13)
  Week 54: number analyzed (Participants) | 346 | 384 | 322
  Week 54 | 0.3 (3.74) | 0.7 (3.69) | 0.8 (4.53)

17. Secondary Outcome: Change From Baseline in Hemoglobin Values
Description: Blood samples of participants were collected for Hemoglobin. Change from baseline in Hemoglobin was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 4, 16, 36 and 48
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 496 | 494 | 489
grams per litre (g/L)
  Week 4: number analyzed (Participants) | 453 | 457 | 457
  Week 4 | -0.4 (6.45) | -2.5 (6.92) | -3.7 (6.19)
  Week 16: number analyzed (Participants) | 423 | 444 | 407
  Week 16 | -0.6 (7.01) | -6.2 (7.76) | -11.9 (8.65)
  Week 36: number analyzed (Participants) | 382 | 398 | 363
  Week 36 | -2.0 (7.25) | -6.4 (8.04) | -12.5 (9.38)
  Week 48: number analyzed (Participants) | 346 | 377 | 334
  Week 48 | -1.9 (7.86) | -6.5 (8.45) | -12.2 (10.62)

18. Secondary Outcome: Change From Baseline in Hematocrit Values
Description: Blood samples of participants were collected for Hematocrit . Change from baseline in Hematocrit was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 4, 8, 12, 16, 36 and 48
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: litre
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 496 | 494 | 489
litre
  Week 4: number analyzed (Participants) | 453 | 457 | 457
  Week 4 | -0.0007 (0.02133) | -0.0068 (0.02189) | -0.0115 (0.01994)
  Week 16: number analyzed (Participants) | 423 | 444 | 407
  Week 16 | -0.0003 (0.02318) | -0.0174 (0.02460) | -0.0339 (0.02697)
  Week 36: number analyzed (Participants) | 382 | 398 | 363
  Week 36 | -0.0037 (0.02246) | -0.0167 (0.02471) | -0.0352 (0.02834)
  Week 48: number analyzed (Participants) | 346 | 377 | 334
  Week 48 | -0.0029 (0.02447) | -0.0177 (0.02658) | -0.0346 (0.03177)

19. Secondary Outcome: Mean Change From Baseline in Short Term Memory Assessment Score
Description: Short term memory assessment score was based on ADAS-Cog questionnaire (Question 1 and 7). ADAS is a performance-based test that measures specific cognitive and behavioral dysfunctions in participants with AD. Question 1 (Word Recall) and Question 7 (Word Recognition) of the ADAS-Cog questionnaire were summed to get a short term memory assessment score. Word recall task consist of the participants score was the mean number of words not recalled on three trials (maximum score 10) and word recognition task, to score this item the number of incorrect responses was counted (maximum error score was 12). The total score ranged from 0 to 22 with 0 indicating absence of symptoms and higher scores indicating greater dysfunction; a negative change from baseline indicated improvement. Change from Baseline in short term memory assessment was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 8, 16, 24, 36, 48 and 56
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  Week 8: number analyzed (Participants) | 430 | 455 | 431
  Week 8 | -0.3 (2.71) | -0.4 (3.03) | -0.3 (2.76)
  Week 16: number analyzed (Participants) | 416 | 433 | 404
  Week 16 | -0.4 (2.93) | -0.7 (2.92) | -0.4 (3.07)
  Week 24: number analyzed (Participants) | 402 | 418 | 377
  Week 24 | 0.1 (2.96) | -0.4 (3.03) | -0.1 (3.06)
  Week 36: number analyzed (Participants) | 372 | 393 | 358
  Week 36 | 0.4 (2.79) | 0.3 (3.18) | 0.7 (3.04)
  Week 48: number analyzed (Participants) | 356 | 383 | 329
  Week 48 | 0.6 (3.01) | 0.3 (3.07) | 0.4 (3.06)
  Week 54: number analyzed (Participants) | 333 | 367 | 305
  Week 54 | 1.1 (2.96) | 0.8 (3.10) | 0.9 (3.17)

20. Secondary Outcome: Change From Baseline in HbA1c at Week 12, Week 24 and Week 36
Description: Blood samples of participants were collected for HbA1c assessment. HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Change from Baseline in HbA1c was calculated as the value at time point minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 12, 24 and 36
Population: Safety population. Week 12, Week 24 and Week 36 assessments of HbA1c were only needed in participants whose HbA1c was >= 6.5% at screening or who had known Type 2 diabetes. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of total hemoglobin
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 145 | 150 | 127
Percent of total hemoglobin
  Week 12: number analyzed (Participants) | 82 | 78 | 81
  Week 12 | 0.01 (0.336) | 0.14 (0.634) | 0.16 (0.407)
  Week 24: number analyzed (Participants) | 145 | 150 | 124
  Week 24 | 0.07 (0.401) | 0.12 (0.422) | 0.06 (0.551)
  Week 36: number analyzed (Participants) | 140 | 145 | 127
  Week 36 | 0.20 (0.400) | 0.19 (0.430) | 0.15 (0.526)

21. Secondary Outcome: Number of Participants With Laboratory Potential Clinical Concern (PCC) Values
Description: Only those parameters for which at least one value of clinical concern (CC) was reported are summarized. Pre-defined limits of potential clinical concern (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) are: Hematocrit 0.8, 1.2; hemoglobin 10-11, 16.5-18; Red blood corpuscles(RBC) 0.8, 1.2; mean corpuscular volume (MCV) 0.8, 1.2; mean corpuscular hemoglobin (MCH) 0.8, 1.2; White blood corpuscles (WBC) 3- absolute value, 15-absolute value, Red Cell Distribution Width (RDW) 0.8, 1.2; Lymphocytes 0.75, 1.5; Monocytes NA, 2; Eosinophil NA, 2; platelet count 100-absolute, 500-absoulte; segmented neutrophil (SN) 0.75, 1.5 and Total Neutrophil (TN) 0.75, 1.5.
Time Frame: Baseline (Week 0), Week 4, 8, 12, 16, 24, 36, 48 and 56
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 496 | 494 | 489
participants
  Eosinophils high: number analyzed (Participants) | 471 | 486 | 477
  Eosinophils high | 0 | 3 | 0
  Hematocrit low: number analyzed (Participants) | 471 | 486 | 477
  Hematocrit low | 2 | 2 | 5
  Hemoglobin high: number analyzed (Participants) | 471 | 486 | 477
  Hemoglobin high | 2 | 0 | 0
  Hemoglobin low: number analyzed (Participants) | 471 | 486 | 477
  Hemoglobin low | 8 | 11 | 31
  Lymphocytes high: number analyzed (Participants) | 471 | 486 | 477
  Lymphocytes high | 0 | 1 | 2
  Lymphocytes low: number analyzed (Participants) | 471 | 486 | 477
  Lymphocytes low | 8 | 10 | 13
  Mean CH high: number analyzed (Participants) | 471 | 486 | 477
  Mean CH high | 0 | 0 | 1
  Mean CH low: number analyzed (Participants) | 471 | 486 | 477
  Mean CH low | 2 | 2 | 0
  Mean CV high: number analyzed (Participants) | 471 | 486 | 477
  Mean CV high | 0 | 0 | 1
  Mean CV low: number analyzed (Participants) | 471 | 486 | 477
  Mean CV low | 2 | 1 | 0
  Monocytes low: number analyzed (Participants) | 471 | 486 | 477
  Monocytes low | 81 | 55 | 65
  Platelet count high: number analyzed (Participants) | 471 | 486 | 475
  Platelet count high | 4 | 2 | 7
  Platelet count low: number analyzed (Participants) | 471 | 486 | 475
  Platelet count low | 1 | 2 | 4
  RDW high: number analyzed (Participants) | 471 | 486 | 475
  RDW high | 18 | 31 | 86
  RBC high: number analyzed (Participants) | 471 | 486 | 477
  RBC high | 0 | 1 | 0
  RBC low: number analyzed (Participants) | 471 | 486 | 477
  RBC low | 0 | 1 | 8
  SN high: number analyzed (Participants) | 471 | 486 | 477
  SN high | 8 | 2 | 4
  SN low: number analyzed (Participants) | 471 | 486 | 477
  SN low | 2 | 6 | 13
  TN high: number analyzed (Participants) | 471 | 486 | 477
  TN high | 4 | 1 | 2
  TN low: number analyzed (Participants) | 471 | 486 | 477
  TN low | 2 | 6 | 13
  WBC high: number analyzed (Participants) | 471 | 486 | 477
  WBC high | 4 | 1 | 3
  WBC low: number analyzed (Participants) | 471 | 486 | 477
  WBC low | 1 | 5 | 12

22. Secondary Outcome: Change From Baseline in Alzheimer's Carer Quality of Life Instrument (ACQLI) Total Score
Description: The ACQLI was an assessment of caregiver quality of life. This instrument consists of 30 questions exploring various aspects of carer's quality of life. Each of the questions had a two point response and the 30 questions were summed to provide a total score. Items are assumed to be unidimensional (i.e., represent a single variable) and are scored 0/1 (false/true) before summation into a total score with a 0-30 range. The total score ranged from 0 to 30, where 0 indicated absence of symptoms and higher score indicated worse outcomes; a negative change from baseline indicated improvement. Change from baseline was calculated as endpoint value minus the baseline value.
Time Frame: Baseline (Week 0), Week 12, 36 and 48
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
Number analyzed (Participants) | 461 | 473 | 459
Score on a scale
  Week 12: number analyzed (Participants) | 387 | 405 | 377
  Week 12 | 0.5 (0.23) | -0.2 (0.23) | -0.0 (0.22)
  Week 36: number analyzed (Participants) | 341 | 363 | 327
  Week 36 | 1.0 (0.28) | 0.6 (0.27) | 0.6 (0.26)
  Week 48: number analyzed (Participants) | 315 | 350 | 309
  Week 48 | 1.2 (0.30) | 0.3 (0.28) | 1.1 (0.31)
Statistical Analysis 1: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — Week 12; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.091, Mixed Models Analysis — Week 12; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis — Week 36; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.3]
Statistical Analysis 4: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis — Week 36; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.4]
Statistical Analysis 5: Comparison: Placebo vs 2mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.6 to -0.1]
Statistical Analysis 6: Comparison: Placebo vs 8mg Rosiglitazone Extended Release; Test type: Superiority or Other; p = 0.797, Mixed Models Analysis — Week 48; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.7]

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: An AE is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug .The data was reported for prospective period. Participants with available data in the prospective period were analysed.
Arm/Group | Placebo | 2mg Rosiglitazone Extended Release | 8mg Rosiglitazone Extended Release
All-Cause Mortality (participants affected / at risk) | 12/496 | 6/494 | 8/489
Serious Adverse Events (participants affected / at risk) | 62/496 | 45/494 | 50/489
Other Adverse Events (participants affected / at risk) | 11/496 | 29/494 | 69/489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=496) | 2mg Rosiglitazone Extended Release (N=494) | 8mg Rosiglitazone Extended Release (N=489)
Hip fracture (Injury, poisoning and procedural complications) | 3 | 4 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of joint (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1 | 6
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lateral patellar compression syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=496) | 2mg Rosiglitazone Extended Release (N=494) | 8mg Rosiglitazone Extended Release (N=489)
Oedema peripheral (General disorders) | 11 | 29 | 69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.